CLINICAL TRIAL: NCT00903331
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter, Parallel Group Study to Evaluate the Efficacy, Safety, and Tolerability of Macitentan in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Macitentan Use in an Idiopathic Pulmonary Fibrosis Clinical Study
Acronym: MUSIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055B201
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; MUSIC
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT-064922 (Experimental): ACT-064922 tablet (macitentan), 10 mg, once daily
  Interventions: Drug: ACT-064992 (macitentan)
- Placebo (Placebo Comparator): Matching placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-064992 (macitentan) — ACT-064992 (macitentan) tablet, 10 mg, once daily
  Other Names: macitentan
  Arms: ACT-064922
Drug: Placebo — matching placebo, once daily
  Arms: Placebo

SUMMARY:
The AC-055B201/MUSIC study is a Phase II study, comparing one dose of ACT-064922 (macitentan) 10 mg with placebo in patients with idiopathic pulmonary fibrosis (IPF). The main study objective is to demonstrate that macitentan positively affects the forced vital capacity (FVC) in comparison with placebo in patients with idiopathic pulmonary fibrosis (IPF).

The secondary objectives are to evaluate the effect of macitentan on the time to disease worsening or death in patients with IPF, and to evaluate the benefit/risk profile of macitentan in the treatment of patients with IPF.

DETAILED DESCRIPTION:
The study included two treatment periods: Period 1 (fixed duration) from randomization up to the primary endpoint evaluation (Month 12 or earlier in case of premature discontinuation of study drug) and Period 2 (variable duration) from the primary endpoint evaluation visit up to the end of study (EOS). EOS occurred when the last patient randomized and not prematurely discontinued completed Period 1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female patients of at least 18 years of age (females of child-bearing potential must use a reliable method of contraception).
3. IPF diagnosis within 3 years prior to randomization, proven according to the American Thoracic Society/European Respiratory Society consensus conference criteria, with surgical lung biopsy.

Exclusion Criteria:

1. Interstitial lung disease due to conditions other than IPF.
2. Presence of extensive honeycombing on Baseline high-resolution computed tomography (HRCT) scan performed within 3 months prior to randomization.
3. Severe concomitant illness limiting life expectancy (< 1 year).
4. Severe restrictive lung disease: forced vital capacity (FVC) < 50% predicted, or FVC < 1.2 liter.
5. Diffusing capacity of the lung for carbon monoxide (DLCO) < 30% predicted.
6. Residual volume ≥ 120% predicted.
7. Obstructive lung disease: forced expiratory volume in 1 second (FEV1)/FVC) < 0.70.
8. Documented sustained improvement of the patient's IPF condition up to 12 months prior to randomization with or without IPF-specific therapy.
9. Recent pulmonary or upper respiratory tract infection (up to 4 weeks prior to randomization).
10. Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements (e.g., pulmonary function tests).
11. Chronic heart failure with New York Heart Association class III/IV or known left ventricular ejection fraction < 25%.
12. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
13. Estimated creatinine clearance < 30 mL/min.
14. Aspartate aminotransferase (AST) and/or alanine aminotransferase > 1.5 x upper limit of normal.
15. Hemoglobin < 75% of the lower limit of the normal range.
16. Systolic blood pressure < 100 mmHg.
17. Pregnant or breast-feeding.
18. Current drug or alcohol dependence.
19. Chronic treatment with the following drugs (within 4 weeks of randomization):

    * Oral corticosteroids (> 20 mg/day of prednisone or equivalent),
    * Immunosuppressive or cytotoxic drugs including cyclophosphamide and azathioprine,
    * Antifibrotic drugs including pirfenidone, D penicillamine, colchicine, tumor necrosis factor α blockers, imatinib and interferon γ,
    * Chronic use of N-acetylcysteine prescribed for IPF (> 600 mg/day).
    * Oral anticoagulants prescribed for IPF.
20. Treatment with endothelin receptor antagonists within 4 weeks prior to randomization.
21. Systemic treatment within 4 weeks prior to randomization with cyclosporine A or tacrolimus, everolimus, sirolimus (calcineurin or mammalian target of rapamycin (mTOR) inhibitors).
22. Treatment with Cytochrome P450 3A inducers within 4 weeks prior to randomization.
23. Known hypersensitivity to drugs of the same class as the study drug, or any of their excipients.
24. Planned treatment, or treatment with another investigational drug within 4 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loic Perchenet, Ph.D., Study Chair — Actelion
Locations (53):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates, P.A., Phoenix, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - U.C. Davis University of California, Sacramento, California
  - UCSD Pulmonary Critical Care, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University Medical Center - Chest Clinic, Stanford, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Wichita Clinic P.A, Wichita, Kansas
  - St. Luke's Medical Group, Chesterfield, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Hospital - Lung Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine - Baylor Clinic, Houston, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (4):
  - Prince Charles Hospital Lung Transplant, Chermside
  - St. Vincent's Public Hospital, Darlinghurst
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Canada (6):
  - University of Alberta - Health Sciences Center, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Hospital Notre-Dame du CHUM, Montreal, Quebec
- France (3):
  - Hopital Avicenne, Bobigny
  - Hôpital Cardiologique et Pneumologique Louis Pradel, Bron
  - CHRU - Hopital Calmette Clinique des Maladies Respiratoires, Lille
- Germany (5):
  - Helios Klinikum Emil von Behring, Berlin
  - Universität zu Köln, Cologne
  - Justus-Liebig-Universität Gießen, Giessen
  - Fachklinik fur Lungenerkrankungen, Immenhausen
  - Ludwig-Maximilian-Universität München, München
- Israel (5):
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petach Tikvah
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Ospedale San Giuseppe Milanocuore, Milan
  - Università degli Studi di Torino Clinica di Malattie dell'Apparato Respiratorio, Orbassano
  - A.O.U Policlinico Tor Vergata, Roma
  - Ospedale di Cattinara, Trieste
- Bolnišnica Golnik, Golnik, Slovenia
- South Africa (2):
  - Centre for Chest Diseases, Milpark Hospital, Johannesburg
  - Pretoria East Hospital, Pretoria
- Spain (5):
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital General Vall d'Hebron, Barcelona
  - Fundación Hospital Alcorcón, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- Karolinska Universitetssjukhuset Lung Allergi kliniken, Stockholm, Sweden
- Turkey (Türkiye) (2):
  - Ankara University School of Medicine, Ankara
  - Ege University School of Medicine, Izmir

REFERENCES:
- [Derived] Raghu G, Million-Rousseau R, Morganti A, Perchenet L, Behr J; MUSIC Study Group. Macitentan for the treatment of idiopathic pulmonary fibrosis: the randomised controlled MUSIC trial. Eur Respir J. 2013 Dec;42(6):1622-32. doi: 10.1183/09031936.00104612. Epub 2013 May 16. PMID 23682110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 48 centers in Australia, Canada, France, Germany, Israel, Italy, Slovenia, South Africa, Spain, Sweden, Turkey, and the USA.
Pre-assignment Details: The study included a screening period of up to 28 days followed by a double-blind treatment phase that was further divided into two periods. 300 patients were screened and 178 randomized in a 2:1 ratio to study treatment with ACT-064922 or placebo
Groups:
- Placebo: Matching placebo, once daily
  Placebo : matching placebo, once daily
- ACT-064922: ACT-064922 tablet, 10 mg, once daily
  ACT-064992 (macitentan) : tablet, 10 mg, once daily
Period: Overall Study
Arm/Group | Placebo | ACT-064922
Started | 59 | 119
Completed | 54 | 101
Not Completed | 5 | 18
Not completed — Death | 4 | 8
Not completed — Withdrawal of consent | 1 | 8
Not completed — Lung transplant | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACT-064922 | Total
Number analyzed (Participants) | 59 | 119 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (6.32) | 65.1 (7.85) | 64.9 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 35 | 57
  Male | 37 | 84 | 121
Region of Enrollment [Number; unit: participants]
  Australia | 9 | 18 | 27
  Canada | 5 | 10 | 15
  France | 10 | 16 | 26
  Germany | 5 | 8 | 13
  Israel | 2 | 5 | 7
  Italy | 1 | 7 | 8
  Slovenia | 1 | 1 | 2
  South Africa | 1 | 1 | 2
  Spain | 4 | 7 | 11
  Sweden | 0 | 1 | 1
  Turkey | 3 | 8 | 11
  United States | 18 | 37 | 55

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC) at Baseline and End of Period 1
Description: FVC was measured at baseline and at the end of Period 1. The same equipment and tester were used during the course of the study. The equipment was calibrated and the calibration documented prior to each patient's measurement. The person responsible for conducting the pulmonary function tests was required to comply with the study guidelines and the American Thoracic Society/European Respiratory Society joint criteria on lung function testing.
Time Frame: 12 months
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: litres
Arm/Group | Placebo | ACT-064922
Number analyzed (Participants) | 59 | 119
litres
  Baseline | 2.74 (0.776) [2.49 to 3.04] | 2.83 (0.834) [2.65 to 3.06]
  End of Period 1 | 2.40 (0.918) [2.10 to 2.70] | 2.57 (1.012) [2.28 to 2.79]
Statistical Analysis 1: Comparison: Placebo vs ACT-064922; The null hypothesis was that there was no difference between ACT-064922 and placebo for the change in FVC from baseline to the end of Period 1. The aim was to detect a placebo-corrected change in FVC of ≥ 0.1 L (Standard Deviation = 0.2 L) at a two-sided 0.05 type 1 error level and 80% power; Test type: Superiority or Other; p = 0.9631, Wilcoxon Rank Sum; Median Difference (Net) = 0.00, 95% CI 2-sided [-0.09 to 0.08]

2. Secondary Outcome: Number of Patients at Risk of Event of Disease Worsening or Death up to the End of Study
Description: Disease worsening was indicated by pulmonary function test/idiopathic pulmonary fibrosis worsening (PFT/IPF) or acute respiratory decompensation of IPF.
  PFT/IPF worsening was indicated by the occurrence of both of the following: confirmed by two tests at least 4 weeks apart, as defined by the occurrence of both of the following: decrease from baseline ≥ 10% in forced vital capacity and decrease from baseline ≥ 15% in corrected diffusing capacity of the lung for carbon monoxide.
  Acute respiratory decompensation of IPF was defined as an unexplained rapid deterioration (over a period of less than 4 weeks) of the patient's condition with increasing shortness of breath requiring oxygen supplementation ≥ 5 L/min to maintain a resting oxygen saturation ≥ 90% or arterial oxygen pressure ≥ 55 mmHg (sea level) or 50 mmHg (high altitude).
Time Frame: Up to end of study (Up to 24 months)
Population: All randomized patients
Measure: Number; unit: participants
Arm/Group | Placebo | ACT-064922
Number analyzed (Participants) | 59 | 119
participants
  Patients at Risk of Event at Month 4 | 59 | 112
  Patients at Risk of Event at Month 8 | 57 | 103
  Patients at Risk of Event at Month 12 | 44 | 81
  Patients at Risk of Event at Month 16 | 22 | 43
  Patients at Risk of Event at Month 20 | 8 | 14
  Patients at Risk of Event at Month 24 | 2 | 1
Statistical Analysis 1: Comparison: Placebo vs ACT-064922; Test type: Superiority or Other; p = 0.7056, Log Rank; Hazard Ratio (HR) = 1.118, 95% CI 2-sided [0.626 to 1.996]

ADVERSE EVENTS:
Time Frame: Up to 28 days after treatment discontinuation, approximately 2 years
Arm/Group | Placebo | ACT-064922
Serious Adverse Events (participants affected / at risk) | 20/59 | 37/119
Other Adverse Events (participants affected / at risk) | 57/59 | 114/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | ACT-064922 (N=119)
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 6 | 10
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 3
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 6
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
COMMUNITY ACQUIRED INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
GASTRIC MUCOSAL HYPERTROPHY (Gastrointestinal disorders) | 0 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
DEVICE MALFUNCTION (General disorders) | 0 | 1
HERNIA OBSTRUCTIVE (General disorders) | 0 | 1
PYREXIA (General disorders) | 0 | 1
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0
SNAKE BITE (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 1 | 0
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT MEDIASTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0
INTESTINAL OPERATION (Surgical and medical procedures) | 0 | 1
MALIGNANT TUMOUR EXCISION (Surgical and medical procedures) | 0 | 1
SKIN LESION EXCISION (Surgical and medical procedures) | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 2 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
WEGENER'S GRANULOMATOSIS (Vascular disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | ACT-064922 (N=119)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 24
COUGH (Respiratory, thoracic and mediastinal disorders) | 21 | 22
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 | 20
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 10 | 17
BRONCHITIS (Infections and infestations) | 9 | 16
OEDEMA PERIPHERAL (General disorders) | 4 | 14
ANAEMIA (Blood and lymphatic system disorders) | 0 | 13
DIZZINESS (Nervous system disorders) | 5 | 11
PULMONARY FUNCTION TEST DECREASED (Investigations) | 5 | 9
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 9
NAUSEA (Gastrointestinal disorders) | 2 | 9
DIARRHOEA (Gastrointestinal disorders) | 5 | 8
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 8
INSOMNIA (Psychiatric disorders) | 3 | 8
HEADACHE (Nervous system disorders) | 8 | 7
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 7
CHEST PAIN (General disorders) | 3 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 6
FATIGUE (General disorders) | 2 | 6
WEIGHT DECREASED (Investigations) | 2 | 6
CONSTIPATION (Gastrointestinal disorders) | 3 | 5
HYPERTENSION (Vascular disorders) | 5 | 4
RASH (Skin and subcutaneous tissue disorders) | 3 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 3
PYREXIA (General disorders) | 5 | 3
ANGINA PECTORIS (Cardiac disorders) | 3 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 | 2
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 3 | 2
ASTHENIA (General disorders) | 4 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 1
VERTIGO (Ear and labyrinth disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less